CLINICAL TRIAL: NCT01779778
Title: The Diurnal and Nocturnal Effect of Travatan With SofZia Preservative on Intraocular Pressure and Ocular Perfusion Pressure
Brief Title: Diurnal and Nocturnal Effect of Travatan With SofZia Preservative on Intraocular Pressure and Ocular Perfusion Pressure
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0175
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to determine the diurnal and nocturnal effects of Travoprost with SofZia (Travatan Z) on intraocular pressure and ocular perfusion pressure.

DETAILED DESCRIPTION:
The investigators hypothesize that Travatan Z will significantly lower intraocular pressure and increase ocular perfusion pressure during both the diurnal and nocturnal period, during a 24-hour evaluation, compared to baseline. The investigators further hypothesize that the medication effects will persist at 72 hours after discontinuation of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma or ocular hypertension, including pigment dispersion glaucoma and pseudoexfoliation glaucoma
* Age ≥ 18 or ≤ 90 years, of either gender, or any race/ethnicity

Exclusion Criteria:

* Females who are currently pregnant or planning to become pregnant, as determined by history during the study period
* Diagnosis of any other form of glaucoma other than open-angle
* Schaffer angle grade < 2 in either eye by gonioscopy
* Chronic, recurrent, or severe inflammatory eye disease
* Intraocular surgery within 6 months or laser within 3 months
* History of active, recurrent, or chronic ocular infection with the Herpes Simplex Virus
* History of cystoid macular edema
* Inability to safely discontinue all ocular medications for 4 weeks
* Patients who smoke or have irregular daily sleep patterns
* Patients who have started or changed glucocorticoids therapy in the last 3 months
* Patients who are currently undergoing medical marijuana therapy
* Any use of a non-FDA approved medication for glaucoma in the last 3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with open angle glaucoma or ocular hypertension
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Changes in Intraocular Pressure | Every 2 hours for 24 hours
  To determine the 24-hour intraocular pressure lowering effect of Travatan Z

SECONDARY OUTCOMES:
Intraocular Pressure Change Duration | 72 hours
  Elucidate the duration of effect from Travatan Z administration which may lead to more efficient dosing regimens

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Seibold, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Eye Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seibold LK, Kahook MY. The diurnal and nocturnal effect of travoprost with sofZia on intraocular pressure and ocular perfusion pressure. Am J Ophthalmol. 2014 Jan;157(1):44-49.e1. doi: 10.1016/j.ajo.2013.09.001. Epub 2013 Oct 30. PMID 24182742